CLINICAL TRIAL: NCT04438577
Title: Evaluation of the Feasibility and Efficacy of Lidocaine Mucilage-ICG as an Optical Agent to Detect Cancer Tissue Delineation During Breast-conserving Surgery
Brief Title: Lidocaine Mucilage-ICG as an Optical Agent for Tumor Delineation During Breast-conserving Surgery
Acronym: LI-CTD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shantou Central Hospital (Other)
Responsible Party: Principal Investigator, Si-Qi Qiu, Principal Investigator, Shantou Central Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ShantouCH
Record Dates: First submitted 2020-06-17; First posted 2020-06-19 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Breast Cancer
Keywords: Breast conserving surgery; fluorescence-guided surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Efficacy of Lidocaine mucilage-ICG (Experimental): Efficacy of Lidocaine mucilage-ICG for intraoperative tumor delineation
  Interventions: Drug: Lidocaine mucilage-ICG

INTERVENTIONS:
Drug: Lidocaine mucilage-ICG — Lidocaine mucilage-ICG as an agent for intraoperative tumor delineation

SUMMARY:
Around 15%-30% of patients receiving breast-conserving surgery (BCS) for invasive breast carcinoma or ductal carcinoma in situ (DCIS) need a reoperation due to tumor-positive margins at final histopathology. Currently available modalities used for intraoperative surgical margin assessment all have specific limitations. In order to improve intraoperative tumor localization and surgical margin assessment in BCS, we developed a fluorescent tracer, the Lidocaine mucilage-ICG tracer, which could be locally injected and detected by fluorescent camera systems during operation. In this study, we aim to evaluate the efficacy of Lidocaine mucilage-ICG as an agent for intraoperative tumor delineation.

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years old
* Histologically or cytologically confirmed breast carcinoma
* Patients planned to receive a breast-conserving surgery
* Patients received a preoperative breast magnetic resonance imaging
* Informed consent form understood and signed
* Patient agrees to all follow-up visits
* Eastern Cooperative Oncology Group(ECOG) performance status 0 to 1 within 14 days of study entry
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the surgery

Exclusion Criteria:

* Psychiatric or other condition that may interfere with the study
* Known allergy or contraindication to any study drug
* Patients received neoadjuvant therapies
* Patients received an excision biopsy of the tumor
* Breast feeding period
* Pregnant (female of childbearing potential only)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Margin width | 7 days
  The distance between tumor and margin on the gross specimen
Positive margin rate | 7 days
  The percentage of patients with a positive margin out of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Si-Qi Qiu, Dr., Principal Investigator — Shantou Central Hospital
Locations (1):
- Shantou Central Hospital, Shantou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No